CLINICAL TRIAL: NCT05295784
Title: Pharmacokinetics (PK) and Safety of Caffeine in Neonates With Hypoxic Ischemic Encephalopathy Receiving Therapeutic Hypothermia
Brief Title: PK and Safety of Caffeine in Neonates With Hypoxic Ischemic Encephalopathy Receiving Therapeutic Hypothermia
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Data no longer support this study
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 260845
Record Dates: First submitted 2022-02-21; First posted 2022-03-25 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-04

CONDITIONS: Acute Kidney Injury; Hypoxic-Ischemic Encephalopathy; Caffeine
MeSH Terms: conditions — Acute Kidney Injury; Hypoxia-Ischemia, Brain | interventions — caffeine citrate

STUDY DESIGN:
Intervention Model Description: Each neonate will receive a single dose of caffeine citrate in the first 24 hours of life. The first six neonates will receive low dose (5 mg/kg), the next six neonates will receive a medium dose (15 mg/kg), and the next six neonates will receive high dose or (25 mg/kg).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Arm 1: Low dose caffeine (Active Comparator): Each neonate will receive a single dose of caffeine citrate in the first 24 hours of life. Arm 1 neonates will receive low dose intravenous caffeine citrate (5 mg/kg).
  Interventions: Drug: Caffeine citrate
- Arm 2: Medium dose caffeine (Active Comparator): Each neonate will receive a single dose of caffeine citrate in the first 24 hours of life. Arm 2 neonates will receive medium dose intravenous caffeine citrate (15 mg/kg).
  Interventions: Drug: Caffeine citrate
- Arm 3: High dose caffeine (Active Comparator): Each neonate will receive a single dose of caffeine citrate in the first 24 hours of life. Arm 3 neonates will receive high dose intravenous caffeine citrate (25 mg/kg).
  Interventions: Drug: Caffeine citrate

INTERVENTIONS:
Drug: Caffeine citrate — A single dose of intravenous caffeine citrate will be administered to neonates with hypoxic ischemic encephalopathy to determine the pharmacokinetics and tolerability.
  Other Names: Cafcit

SUMMARY:
A phase 1 study investigating the tolerability and pharmacokinetics of caffeine citrate in neonates with hypoxic ischemic encephalopathy receiving therapeutic hypothermia. This study is an essential first step to develop caffeine as a kidney protective medication in this in this vulnerable group of newborns.

DETAILED DESCRIPTION:
Neonatal acute kidney injury (AKI) is an unfortunate comorbidity in neonates with hypoxic ischemic encephalopathy (HIE) which is brain injury due to a lack of blood flow and oxygen delivery to a neonate around the time of delivery. Neonatal AKI increases the risk of death by 4 fold. AKI in neonates with HIE is associated with brain injury on brain MRI and worse neurodevelopmental outcomes at 2 years. Despite the increases in death and morbidity associated with AKI, limited therapeutic interventions currently exist.

Caffeine is a promising medication for kidney protection in neonates at high risk for AKI. Three retrospective studies in premature neonates identified a reduction in AKI in neonates exposed to caffeine. Theophylline, which is in the same drug class as caffeine, has been shown to improve urine output and decrease AKI in neonates with HIE. Limited centers worldwide utilize theophylline in neonates with HIE due to its side effects. Caffeine is a well-tolerated and is extensively utilized in neonatal intensive care units (NICUs) in the premature population for prevention of chronic lung disease and for apnea of prematurity (or immature breathing patterns). Therefore, dosing guidelines are well established for preterm neonates and neonatologists are comfortable administering the drug.

Specific Aim 1: Determine the pharmacokinetics (how an organism affects a drug) of caffeine in neonates ≥ 35 weeks GA with HIE receiving therapeutic hypothermia.

Specific Aim 2: Assess the preliminary safety and tolerability of caffeine in neonates with HIE receiving hypothermia including any impact on seizure burden.

Specific Aim 1: Characterize acute kidney injury (AKI) in neonates with HIE receiving therapeutic hypothermia with caffeine exposure using serum creatinine (SCr), urine output, renal near infrared spectroscopy (NIRS), and urinary biomarkers.

General Experimental Approach:

A total of 18 neonates will be enrolled over approximately 18 months. Each neonate will receive a single dose of caffeine in the first 24 hours of life. The first six neonates will receive low dose (5 mg/kg), the next six neonates will receive a medium dose (15 mg/kg), and the next six neonates will receive high dose or (25 mg/kg).

Demographic data (birthdate, sex, ethnicity, race, gestational age) and clinical data (perinatal birth history, other diagnosis) will be collected from the electronic medical record input into a secure REDCap database created uniquely for this study. Laboratory (serum creatinine) and imaging (head ultrasound and brain MRIs) results will also be recorded.

Blood samples will be obtained from the newborns to monitor the caffeine blood levels. Urine samples will be analyzed for biomarkers that detect kidney damage. Data on seizures and medications will be monitored closely. Blood flow and oxygen levels in the kidney will be monitored with a non-invasive technology called near infrared spectroscopy or NIRS. Data will be collected on urine output and blood creatinine levels to determine which newborns have acute kidney injury.

In conclusion, this study will investigate the drug levels in the blood of caffeine in neonates with HIE receiving therapeutic hypothermia. Safety will also be monitored obtained. The investigators anticipate caffeine is a safe and effective therapy. This study is an essential first step to develop caffeine as a kidney protective medication in this in this vulnerable group of newborns.

ELIGIBILITY:
Inclusion Criteria:

1. Newborns ≥ 35 weeks GA
2. Admitted to the ACH NICU less than 24 hours of life
3. Receiving active or passive TH or whole-body cooling at 12 hours of life to treat hypoxic ischemic encephalopathy per institutional criteria based on National Institute of Child Health and Human Development criteria

Exclusion Criteria:

1. Genetic or congenital condition that affects renal function (e.g., congenital anomalies of the kidney and urinary tract (CAKUT), complex congenital heart disease)
2. Diminished capacity or autonomy of the neonate's parents that prevents their ability to give informed consent
3. Theophylline, aminophylline, or caffeine exposure prior to enrollment
4. Status epilepticus as defined by:

   1. A seizure lasting longer than 30 minutes
   2. Use of a continuous infusion of antiepileptic medication (i.e., midazolam)
   3. The use of 3 or more antiepileptic medications for the indications of intractable seizures

Ages: 0 Hours to 24 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2024-05-08 (Actual); Primary Completion 2024-05-08 (Actual); Study Completion 2024-05-08 (Actual)

PRIMARY OUTCOMES:
Clearance of caffeine | 1 week
  Clearance (mL h-1 kg-1)
Volume of distribution of caffeine | 1 week
  Volume of distribution (ml/kg)
Peak plasma concentration (Cmax) of caffeine | 1 week
  Peak plasma concentration (Cmax) (ng/mL)
Area under the plasma concentration-time curve of caffeine | 1 week
  Area under the plasma concentration-time curve from 0 to infinity (AUC0-INF) (mg*h/L)
Seizure incidence | 2 weeks
  Number of neonates who developed seizures based on continuous video electroencephalogram (VEEG) data
Seizure burden | 2 weeks
  Electrographic seizures (in minutes per hour) based on continuous video electroencephalogram (VEEG) data

SECONDARY OUTCOMES:
Acute kidney injury | 10 days
  AKI incidence utilizing KDIGO criteria based on urine output and SCr.
Renal near infrared spectroscopy (NIRS) | 5 days
  Investigate changes in renal NIRS values during the therapeutic hypothermia and rewarming period.
Urine neutrophil gelatinase-associated lipocalin (NGAL) (ng/mL) | 3 days
  Urine samples will be collected at 24, 48 and 72 hours after birth. Urine will be analyzed for NGAL.
Urine kidney injury molecule-1 (KIM-1) (pg/mL) | 3 days
  Urine samples will be collected at 24, 48 and 72 hours after birth. Urine will be analyzed for KIM-1.
Urine interleukin-18 (IL-18) (pg/mL) | 3 days
  Urine samples will be collected at 24, 48 and 72 hours after birth. Urine will be analyzed for IL-18.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Rumpel, MD, Principal Investigator — University of Arkansas
Locations (2):
- United States (2):
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rumpel J, Spray BJ, Chock VY, Kirkley MJ, Slagle CL, Frymoyer A, Cho SH, Gist KM, Blaszak R, Poindexter B, Courtney SE. Urine Biomarkers for the Assessment of Acute Kidney Injury in Neonates with Hypoxic Ischemic Encephalopathy Receiving Therapeutic Hypothermia. J Pediatr. 2022 Feb;241:133-140.e3. doi: 10.1016/j.jpeds.2021.08.090. Epub 2021 Sep 20. PMID 34547334
- [Background] Selewski DT, Jordan BK, Askenazi DJ, Dechert RE, Sarkar S. Acute kidney injury in asphyxiated newborns treated with therapeutic hypothermia. J Pediatr. 2013 Apr;162(4):725-729.e1. doi: 10.1016/j.jpeds.2012.10.002. Epub 2012 Nov 10. PMID 23149172
- [Background] Kirkley MJ, Boohaker L, Griffin R, Soranno DE, Gien J, Askenazi D, Gist KM; Neonatal Kidney Collaborative (NKC). Acute kidney injury in neonatal encephalopathy: an evaluation of the AWAKEN database. Pediatr Nephrol. 2019 Jan;34(1):169-176. doi: 10.1007/s00467-018-4068-2. Epub 2018 Aug 28. PMID 30155763
- [Background] Jetton JG, Boohaker LJ, Sethi SK, Wazir S, Rohatgi S, Soranno DE, Chishti AS, Woroniecki R, Mammen C, Swanson JR, Sridhar S, Wong CS, Kupferman JC, Griffin RL, Askenazi DJ; Neonatal Kidney Collaborative (NKC). Incidence and outcomes of neonatal acute kidney injury (AWAKEN): a multicentre, multinational, observational cohort study. Lancet Child Adolesc Health. 2017 Nov;1(3):184-194. doi: 10.1016/S2352-4642(17)30069-X. PMID 29732396
- [Background] Cavallin F, Rubin G, Vidal E, Cainelli E, Bonadies L, Suppiej A, Trevisanuto D. Prognostic role of acute kidney injury on long-term outcome in infants with hypoxic-ischemic encephalopathy. Pediatr Nephrol. 2020 Mar;35(3):477-483. doi: 10.1007/s00467-019-04406-4. Epub 2019 Dec 11. PMID 31828471
- [Background] Bhatt GC, Gogia P, Bitzan M, Das RR. Theophylline and aminophylline for prevention of acute kidney injury in neonates and children: a systematic review. Arch Dis Child. 2019 Jul;104(7):670-679. doi: 10.1136/archdischild-2018-315805. Epub 2019 Feb 23. PMID 30798259
- [Background] Chock VY, Cho SH, Frymoyer A. Aminophylline for renal protection in neonatal hypoxic-ischemic encephalopathy in the era of therapeutic hypothermia. Pediatr Res. 2021 Mar;89(4):974-980. doi: 10.1038/s41390-020-0999-y. Epub 2020 Jun 5. PMID 32503030
- [Background] Harer MW, Askenazi DJ, Boohaker LJ, Carmody JB, Griffin RL, Guillet R, Selewski DT, Swanson JR, Charlton JR; Neonatal Kidney Collaborative (NKC). Association Between Early Caffeine Citrate Administration and Risk of Acute Kidney Injury in Preterm Neonates: Results From the AWAKEN Study. JAMA Pediatr. 2018 Jun 4;172(6):e180322. doi: 10.1001/jamapediatrics.2018.0322. Epub 2018 Jun 4. PMID 29610830
- [Background] Aviles-Otero N, Kumar R, Khalsa DD, Green G, Carmody JB. Caffeine exposure and acute kidney injury in premature infants with necrotizing enterocolitis and spontaneous intestinal perforation. Pediatr Nephrol. 2019 Apr;34(4):729-736. doi: 10.1007/s00467-018-4140-y. Epub 2018 Nov 10. PMID 30415418
- [Background] Carmody JB, Harer MW, Denotti AR, Swanson JR, Charlton JR. Caffeine Exposure and Risk of Acute Kidney Injury in a Retrospective Cohort of Very Low Birth Weight Neonates. J Pediatr. 2016 May;172:63-68.e1. doi: 10.1016/j.jpeds.2016.01.051. Epub 2016 Feb 18. PMID 26898806
- [Background] AlGadeeb K, Qaraqei M, Algadeeb R, Faqeehi H, Al-Matary A. Prediction of risk factors and outcomes of neonatal acute kidney injury. J Nephrol. 2021 Oct;34(5):1659-1668. doi: 10.1007/s40620-021-01130-x. Epub 2021 Sep 1. PMID 34468977
- [Background] Dobson NR, Patel RM, Smith PB, Kuehn DR, Clark J, Vyas-Read S, Herring A, Laughon MM, Carlton D, Hunt CE. Trends in caffeine use and association between clinical outcomes and timing of therapy in very low birth weight infants. J Pediatr. 2014 May;164(5):992-998.e3. doi: 10.1016/j.jpeds.2013.12.025. Epub 2014 Jan 23. PMID 24461786
- [Background] Lee TC, Charles B, Steer P, Flenady V, Shearman A. Population pharmacokinetics of intravenous caffeine in neonates with apnea of prematurity. Clin Pharmacol Ther. 1997 Jun;61(6):628-40. doi: 10.1016/S0009-9236(97)90097-7. PMID 9209245
- [Background] Charles BG, Townsend SR, Steer PA, Flenady VJ, Gray PH, Shearman A. Caffeine citrate treatment for extremely premature infants with apnea: population pharmacokinetics, absolute bioavailability, and implications for therapeutic drug monitoring. Ther Drug Monit. 2008 Dec;30(6):709-16. doi: 10.1097/FTD.0b013e3181898b6f. PMID 19057373
- [Background] Falcao AC, Fernandez de Gatta MM, Delgado Iribarnegaray MF, Santos Buelga D, Garcia MJ, Dominguez-Gil A, Lanao JM. Population pharmacokinetics of caffeine in premature neonates. Eur J Clin Pharmacol. 1997;52(3):211-7. doi: 10.1007/s002280050276. PMID 9218928
- [Background] Thomson AH, Kerr S, Wright S. Population pharmacokinetics of caffeine in neonates and young infants. Ther Drug Monit. 1996 Jun;18(3):245-53. doi: 10.1097/00007691-199606000-00005. PMID 8738763
- [Background] CAFCIT (caffeine citrate) Injection, CAFCIT (caffeine citrate) Oral solution, Package insert. Available at: https://www.accessdata.fda.gov/drugsatfda_docs/label/2000/20793s1lbl.pdf. Accessed October 30, 2021.
- [Background] Gillot I, Gouyon JB, Guignard JP. Renal effects of caffeine in preterm infants. Biol Neonate. 1990;58(3):133-6. doi: 10.1159/000243252. PMID 2279048
- [Background] Zappitelli M, Ambalavanan N, Askenazi DJ, Moxey-Mims MM, Kimmel PL, Star RA, Abitbol CL, Brophy PD, Hidalgo G, Hanna M, Morgan CM, Raju TNK, Ray P, Reyes-Bou Z, Roushdi A, Goldstein SL. Developing a neonatal acute kidney injury research definition: a report from the NIDDK neonatal AKI workshop. Pediatr Res. 2017 Oct;82(4):569-573. doi: 10.1038/pr.2017.136. Epub 2017 Jul 11. No abstract available. PMID 28604760
- [Background] Echeverri D, Montes FR, Cabrera M, Galan A, Prieto A. Caffeine's Vascular Mechanisms of Action. Int J Vasc Med. 2010;2010:834060. doi: 10.1155/2010/834060. Epub 2010 Aug 25. PMID 21188209
- [Background] Aranda JV, Collinge JM, Zinman R, Watters G. Maturation of caffeine elimination in infancy. Arch Dis Child. 1979 Dec;54(12):946-9. doi: 10.1136/adc.54.12.946. PMID 533298
- [Background] Aranda JV, Beharry KD. Pharmacokinetics, pharmacodynamics and metabolism of caffeine in newborns. Semin Fetal Neonatal Med. 2020 Dec;25(6):101183. doi: 10.1016/j.siny.2020.101183. Epub 2020 Nov 26. PMID 33293242
- [Background] Zanelli S, Buck M, Fairchild K. Physiologic and pharmacologic considerations for hypothermia therapy in neonates. J Perinatol. 2011 Jun;31(6):377-86. doi: 10.1038/jp.2010.146. Epub 2010 Dec 23. PMID 21183927
- [Background] Schmidt B, Roberts RS, Davis P, Doyle LW, Barrington KJ, Ohlsson A, Solimano A, Tin W; Caffeine for Apnea of Prematurity Trial Group. Caffeine therapy for apnea of prematurity. N Engl J Med. 2006 May 18;354(20):2112-21. doi: 10.1056/NEJMoa054065. PMID 16707748
- [Background] Frymoyer A, Van Meurs KP, Drover DR, Klawitter J, Christians U, Chock VY. Theophylline dosing and pharmacokinetics for renal protection in neonates with hypoxic-ischemic encephalopathy undergoing therapeutic hypothermia. Pediatr Res. 2020 Dec;88(6):871-877. doi: 10.1038/s41390-020-01140-8. Epub 2020 Sep 12. PMID 32919393
- [Background] Schmidt B, Roberts RS, Davis P, Doyle LW, Barrington KJ, Ohlsson A, Solimano A, Tin W; Caffeine for Apnea of Prematurity Trial Group. Long-term effects of caffeine therapy for apnea of prematurity. N Engl J Med. 2007 Nov 8;357(19):1893-902. doi: 10.1056/NEJMoa073679. PMID 17989382
- [Background] Schmidt B, Anderson PJ, Doyle LW, Dewey D, Grunau RE, Asztalos EV, Davis PG, Tin W, Moddemann D, Solimano A, Ohlsson A, Barrington KJ, Roberts RS; Caffeine for Apnea of Prematurity (CAP) Trial Investigators. Survival without disability to age 5 years after neonatal caffeine therapy for apnea of prematurity. JAMA. 2012 Jan 18;307(3):275-82. doi: 10.1001/jama.2011.2024. PMID 22253394
- [Background] Schmidt B, Roberts RS, Anderson PJ, Asztalos EV, Costantini L, Davis PG, Dewey D, D'Ilario J, Doyle LW, Grunau RE, Moddemann D, Nelson H, Ohlsson A, Solimano A, Tin W; Caffeine for Apnea of Prematurity (CAP) Trial Group. Academic Performance, Motor Function, and Behavior 11 Years After Neonatal Caffeine Citrate Therapy for Apnea of Prematurity: An 11-Year Follow-up of the CAP Randomized Clinical Trial. JAMA Pediatr. 2017 Jun 1;171(6):564-572. doi: 10.1001/jamapediatrics.2017.0238. PMID 28437520
- [Background] McPherson C, Neil JJ, Tjoeng TH, Pineda R, Inder TE. A pilot randomized trial of high-dose caffeine therapy in preterm infants. Pediatr Res. 2015 Aug;78(2):198-204. doi: 10.1038/pr.2015.72. Epub 2015 Apr 9. PMID 25856169
- [Background] Vesoulis ZA, McPherson C, Neil JJ, Mathur AM, Inder TE. Early High-Dose Caffeine Increases Seizure Burden in Extremely Preterm Neonates: A Preliminary Study. J Caffeine Res. 2016 Sep 1;6(3):101-107. doi: 10.1089/jcr.2016.0012. PMID 27679737
- [Background] Chock VY, Frymoyer A, Yeh CG, Van Meurs KP. Renal Saturation and Acute Kidney Injury in Neonates with Hypoxic Ischemic Encephalopathy Undergoing Therapeutic Hypothermia. J Pediatr. 2018 Sep;200:232-239.e1. doi: 10.1016/j.jpeds.2018.04.076. Epub 2018 Jun 1. PMID 29866591
- [Background] Perera V, Gross AS, McLachlan AJ. Caffeine and paraxanthine HPLC assay for CYP1A2 phenotype assessment using saliva and plasma. Biomed Chromatogr. 2010 Oct;24(10):1136-44. doi: 10.1002/bmc.1419. PMID 20853468
- [Background] Lynch NE, Stevenson NJ, Livingstone V, Mathieson S, Murphy BP, Rennie JM, Boylan GB. The temporal characteristics of seizures in neonatal hypoxic ischemic encephalopathy treated with hypothermia. Seizure. 2015 Dec;33:60-5. doi: 10.1016/j.seizure.2015.10.007. Epub 2015 Oct 23. PMID 26571073